CLINICAL TRIAL: NCT05523843
Title: Pilot Study on the Clinical Utility of the Tulsa Life Chart: A Graphical Representation of Patient Life History
Brief Title: Pilot Study on the Clinical Utility of the Tulsa Life Chart
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Principal Investigator, Robin Aupperle, Principal Investigator, Laureate Institute for Brain Research, Inc.
Other Study IDs: 2022-004
Record Dates: First submitted 2022-08-22; First posted 2022-08-31 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Mental Health Issue; Mental Health Disorder; Assessment, Self
Keywords: Assessment; Life Chart; Web-based application; Clinical intake assessment; Pragmatic Clinical Pilot
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment seeking individuals: Individuals seeking treatment in the Laureate Psychiatric Clinic and Hospital (LPCH).
  Interventions: Other: Tulsa Life Chart (TLC)
- Healthcare professionals: Healthcare professionals (HCPS) include nurses, psychologists, therapists, medical doctors, dieticians, etc who work at LPCH and are engaged in direct patient care.

INTERVENTIONS:
Other: Tulsa Life Chart (TLC) — The TLC is a self-administered, interactive assessment of patient history. Participants are asked to provide information from birth to their current age in developmental epochs (i.e., ages 0 to 5; 6 to 10; 11 to 14; 15 to 18; 19 to 25; 26 to 35; and so on in 10-year increments). Participants are first asked to rate their average mood during the epoch. They are then asked about locations lived, schools attended, people they were close to, hobbies, medical conditions, medications, hospitalizations, direct and indirect substance use exposure, mental health symptoms, mental health treatment, and important life events. The information is then displayed in an interactive, graphic of the individual's life that is reviewable by the patient and the healthcare providers enrolled in the study that the patient consents to having access.
  Groups: Treatment seeking individuals

SUMMARY:
The proposed study aims to examine the usability, utility, and feasibility of the Tulsa Life Chart (TLC) in a sample of patients seeking mental health treatment and their healthcare providers. The TLC is an interactive, web-based application used to create a graphical interface for visualizing a patient's life history.

DETAILED DESCRIPTION:
Understanding the longitudinal course of mental health is critical for case conceptualization. One approach for capturing the complexity of an individual's illness course is to depict it graphically. The first attempt for this method was the National Institute of Mental Health Life Chart for Bipolar Disorder. Subsequent research indicated Life Charts are useful clinically and time- and cost-effective. Despite clinical utility and time and cost efficiency, this approach has not been widely adopted in the mental health field. Possible explanations are the prior focus on bipolar disorder, time required to collect information, and prior versions have not had automatic translation of the patient information into an image.

The Tulsa Life Chart (TLC) was developed by researchers at the Laureate Institute for Brain Research (LIBR). The TLC was developed to address weaknesses of previous life chart methods and help patients and healthcare professionals (HCPs) quickly identify patterns of mental health symptoms across diagnostic categories. To date only one formal exploration of the TLC has been conducted in a sample of individuals with mood, anxiety, eating disorders, and substance use disorders, which suggested that participants felt the TLC was helpful in understanding their mental health symptoms and was pleasant to complete. Unpublished focus groups with HCPs suggest HCPs believe the TLC could help to improve patient encounters by increasing understanding of patients and facilitating conversations. Based on these findings the goal of the proposed study is to examine clinical usability, utility, and feasibility in a pragmatic pilot trial.

The current trial will recruit individuals seeking treatment within the Laureate Psychiatric Clinic and Hospital and healthcare professionals involved with their care. Treatment-seeking patients who are invited to participate will be asked to complete the TLC soon after establishing care in a health system setting. Subsequently, the patient's HCP will review the chart during the intake process and complete several measures related to the chart and their experience (baseline assessment point). Patients and HCPs will engage in treatment as usual in between the TLC and assessment time points. Prior to or shortly following discharge/termination of treatment (approximately 4 to 12 weeks depending on the clinic), patients and HCPs will be asked to again complete questions to determine the TLC's usefulness during treatment. The overarching aim of the current study is to examine the usefulness of the Tulsa Life Chart for treatment-seeking individuals and healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

Treatment Seekers Inclusion Criteria:

1. Actively seeking mental health treatment at Laureate Psychiatric Clinic and Hospital
2. Provision of informed consent or if <18 assent and parental consent
3. Age 15 to 65 years
4. Necessary resources to engage in a technology-based intervention
5. English proficiency
6. Willingness to grant access to medical records

HCPs Inclusion Criteria:

1. Employed at Laureate Psychiatric Clinic and Hospital in a patient care role
2. Informed consent
3. English proficiency
4. Access to resources to engage in technology-based intervention

Exclusion Criteria:

Treatment Seekers Exclusion Criteria:

1. Active suicidal ideation with plan or intent
2. No access to resources to participate in a technology-based intervention
3. Completed more than 2 sessions of therapy with their current provider prior to enrollment in the study
4. Not proficient in English

HCPs Exclusion Criteria:

1. No access to resources to participate in a technology-based intervention
2. Not proficient in English

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Indviduals seeking mental health treatment and their healthcare providers who have been invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
mHealth App Usability Questionnaire (MAUQ) Total Usability Score (Patient) | Baseline assessment
  Validated self-report survey in which participants indicate how usable the assessment tool was, with scores ranging from 18 to 126. Higher scores indicate greater usability.
mHealth App Usability Questionnaire (MAUQ) Total Usability Score (Healthcare Professional) | Baseline assessment
  Validated self-report survey in which healthcare professional participants indicate how usable the assessment tool was, with scores ranging from 18 to 126. Higher scores indicate greater usability.

SECONDARY OUTCOMES:
mHealth App Usability Questionnaire (MAUQ) - Ease of Use Subscale (Patient) | Baseline assessment
  Subscale of a validated self-report survey in which patient participants report how easy the assessment tool was to use. Ease of use scores range from 5 to 35 with higher scores indicating greater ease of use.
mHealth App Usability Questionnaire (MAUQ) - Ease of Use Subscale (Healthcare Professional) | Baseline assessment
  Subscale of a validated self-report survey in which healthcare professional participants report how easy the assessment tool was to use. Ease of use scores range from 5 to 35 with higher scores indicating greater ease of use.
mHealth App Usability Questionnaire (MAUQ) - Interface and Satisfaction Subscale (Patient) | Baseline assessment
  Subscale of a validated self-report survey in which patients rate their satisfaction with the assessment tool and the interface of the tool. Interface and satisfaction scores range from 7 to 49 with higher scores indicating greater satisfaction.
mHealth App Usability Questionnaire (MAUQ) - Interface and Satisfaction Subscale (Healthcare Professional) | Baseline assessment
  Subscale of a validated self-report survey in which healthcare professionals rate their satisfaction with the assessment tool and the interface of the tool. Interface and satisfaction scores range from 7 to 49 with higher scores indicating greater satisfaction.
mHealth App Usability Questionnaire (MAUQ) - Usefulness Subscale (Patient) | Baseline assessment
  Subscale of a validated self-report survey in which patients rate the usefulness of the assessment tool. Usefulness scores range from 6 to 42 with higher scores indicating greater usefulness.
mHealth App Usability Questionnaire (MAUQ) - Usefulness Subscale (Healthcare Professional) | Baseline assessment
  Subscale of a validated self-report survey in which healthcare professionals rate the usefulness of the assessment tool. Usefulness scores range from 6 to 42 with higher scores indicating greater usefulness.
Time spent to complete the Tulsa Life Chart (Patient) | Baseline assessment
  Treatment seekers self-report of time to complete the TLC and embedded time count from the TLC application.
Time spent to reviewing the Tulsa Life Chart (Healthcare Professional) | Baseline assessment
  Healthcare professionals' self-report of time spent reviewing the TLC and embedded time count from the TLC application.

OTHER OUTCOMES:
mHealth App Usability Questionnaire (MAUQ) Total Usability Score (Patient) | Assessment two - on average 4 to 12 weeks after baseline assessment
  Validated self-report survey in which participants indicate how usable the assessment tool was, with scores ranging from 18 to 126. Higher scores indicate greater usability.
Change in perception of usefulness | Change from baseline to the post-treatment timepoint, approximately 4 - 12 weeks after baseline
  Change in mHealth App Usability Questionnaire (MAUQ) score from first assessment time point to second assessment time point. Scores on the MAUQ range from 18 to 126. Higher scores indicate greater usability.
mHealth App Usability Questionnaire (MAUQ) - Ease of Use Subscale (Patient) | Assessment two - on average 4 to 12 weeks after baseline assessment
  Subscale of a validated self-report survey in which patient participants report how easy the assessment tool was to use. Ease of use scores range from 5 to 35 with higher scores indicating greater ease of use.
mHealth App Usability Questionnaire (MAUQ) - Ease of Use Subscale (Healthcare Professional) | Assessment two - on average 4 to 12 weeks after baseline assessment
  Subscale of a validated self-report survey in which healthcare professional participants report how easy the assessment tool was to use. Ease of use scores range from 5 to 35 with higher scores indicating greater ease of use.
mHealth App Usability Questionnaire (MAUQ) - Interface and Satisfaction Subscale (Patient) | Assessment two - on average 4 to 12 weeks after baseline assessment
  Subscale of a validated self-report survey in which patients rate their satisfaction with the assessment tool and the interface of the tool. Interface and satisfaction scores range from 7 to 49 with higher scores indicating greater satisfaction.
mHealth App Usability Questionnaire (MAUQ) - Interface and Satisfaction Subscale (Healthcare Professional) | Assessment two - on average 4 to 12 weeks after baseline assessment
  Subscale of a validated self-report survey in which healthcare professionals rate their satisfaction with the assessment tool and the interface of the tool. Interface and satisfaction scores range from 7 to 49 with higher scores indicating greater satisfaction.
mHealth App Usability Questionnaire (MAUQ) - Usefulness Subscale (Patient) | Assessment two - on average 4 to 12 weeks after baseline assessment
  Subscale of a validated self-report survey in which patients rate the usefulness of the assessment tool. Usefulness scores range from 6 to 42 with higher scores indicating greater usefulness.
mHealth App mHealth App Usability Questionnaire (MAUQ) - Usefulness Subscale (Healthcare Professional) | Assessment two - on average 4 to 12 weeks after baseline assessment
  Subscale of a validated self-report survey in which healthcare professionals rate the usefulness of the assessment tool. Usefulness scores range from 6 to 42 with higher scores indicating greater usefulness.
Utility Questionnaire (Patient) | Baseline assessment
  This measure was created for the purpose of the current study to measure how useful the assessment tool was in multiple domains. This measure asks treatment seekers questions pertaining to their experience using the Tulsa Life Chart including: ease of understanding and impact of completing the Tulsa Life Chart on remembering life events, understanding of mental health patterns, communication with their provider, and motivation for treatment engagement. Scores range from 6 to 28 with higher scores indicating greater utility for patients.
Utility Questionnaire (Healthcare Professional) | Baseline assessment
  This measure was created for the purpose of the current study to measure how useful the assessment tool was in multiple domains. This measure asks healthcare professionals questions pertaining to their experience viewing their patient's Tulsa Life Chart. Domains include ease of understanding the chart; usefulness in diagnosing their patient; and impact on understanding patient's psychosocial history, understanding patterns in their patient's mental health, and facilitating conversations. Scores range from 7 to 35 with higher scores indicating greater utility for healthcare professionals.
Utility Questionnaire (Patient) | Assessment two - on average 4 to 12 weeks after baseline assessment
  This measure was created for the purpose of the current study to measure how useful the assessment tool was in multiple domains. This measure asks treatment seekers questions pertaining to their experience using the Tulsa Life Chart including: ease of understanding and impact of completing the Tulsa Life Chart on remembering life events, understanding of mental health patterns, communication with their provider, and motivation for treatment engagement. Scores range from 5 to 23 with higher scores indicating greater utility for patients.
Utility Questionnaire (Healthcare Professional) | Assessment two - on average 4 to 12 weeks after baseline assessment
  This measure was created for the purpose of the current study to measure how useful the assessment tool was in multiple domains. This measure asks healthcare professionals questions pertaining to their experience viewing their patient's Tulsa Life Chart. Domains include impact on therapy; ease of understanding the chart; usefulness in diagnosing their patient; and impact on understanding patient's psychosocial history, understanding patterns in their patient's mental health, and facilitating conversations. Scores range from 8 to 35 with higher scores indicating greater utility for healthcare professionals.
Likelihood of recommending the Tulsa Life Chart to other patients (Patient) | Baseline assessment
  One question will be used to assess the patient's likelihood of recommending the Tulsa Life Chart. "How likely are you to recommend the Tulsa Life Chart to someone else who may be experiencing mental health symptoms?" Scores range from 1 to 5, with higher scores indicating greater likelihood of recommending to the chart.
Likelihood of recommending the Tulsa Life Chart to other healthcare professionals (Healthcare Professional) | Baseline assessment
  One question will be used to assess the patient's likelihood of recommending the Tulsa Life Chart to other healthcare professionals. "Based on this experience, how likely are you to recommend the Tulsa Life Chart to other providers?" Scores range from 1 to 5, with higher scores indicating greater likelihood of recommending to the chart.
Likelihood of recommending the Tulsa Life Chart to other patients (Patient) | Assessment two - on average 4 to 12 weeks after baseline assessment
  One question will be used to assess the patient's likelihood of recommending the Tulsa Life Chart. "How likely are you to recommend the Tulsa Life Chart to someone else who may be experiencing mental health symptoms?" Scores range from 1 to 5, with higher scores indicating greater likelihood of recommending to the chart.
Likelihood of recommending (Healthcare Professional) | Assessment two - on average 4 to 12 weeks after baseline assessment
  One question will be used to assess the patient's likelihood of recommending the Tulsa Life Chart to other healthcare professionals. "Based on this experience, how likely are you to recommend the Tulsa Life Chart to other providers?" Scores range from 1 to 5, with higher scores indicating greater likelihood of recommending to the chart.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Aupperle, PhD, Principal Investigator — Laureate Institute for Brain Research
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
The current study is enrolling participants from a specific treatment center and the data being collected and visualized as part fo the Tulsa Life Chart would be able to be used to potentially identify the individual participants. Thus, no data from this study will be shared through open access databases. If the visualization data from the TLC is shared for publication, data will be modified to for participant confidentiality and privacy. Data obtained from questionnaire measures may be shared upon request.

REFERENCES:
- [Background] Aupperle RL, Paulus MP, Kuplicki R, Touthang J, Victor T, Yeh HW; Tulsa 1000 Investigators; Khalsa SS. Web-Based Graphic Representation of the Life Course of Mental Health: Cross-Sectional Study Across the Spectrum of Mood, Anxiety, Eating, and Substance Use Disorders. JMIR Ment Health. 2020 Jan 28;7(1):e16919. doi: 10.2196/16919. PMID 32012081
- [Background] Manderscheid RW, Ryff CD, Freeman EJ, McKnight-Eily LR, Dhingra S, Strine TW. Evolving definitions of mental illness and wellness. Prev Chronic Dis. 2010 Jan;7(1):A19. Epub 2009 Dec 15. PMID 20040234
- [Background] Post RM, Roy-Byrne PP, Uhde TW. Graphic representation of the life course of illness in patients with affective disorder. Am J Psychiatry. 1988 Jul;145(7):844-8. doi: 10.1176/ajp.145.7.844. PMID 3381929
- [Background] Born C, Amann BL, Grunze H, Post RM, Scharer L. Saving time and money: a validation of the self ratings on the prospective NIMH Life-Chart Method (NIMH-LCM). BMC Psychiatry. 2014 May 7;14:130. doi: 10.1186/1471-244X-14-130. PMID 24886463
- [Background] Denicoff KD, Ali SO, Sollinger AB, Smith-Jackson EE, Leverich GS, Post RM. Utility of the daily prospective National Institute of Mental Health Life-Chart Method (NIMH-LCM-p) ratings in clinical trials of bipolar disorder. Depress Anxiety. 2002;15(1):1-9. doi: 10.1002/da.1078. PMID 11816046